CLINICAL TRIAL: NCT03270397
Title: Addressing Body Image Issues While Teaching Academic Course: Efficacy Trial of Innovative Academic Initiative
Brief Title: Addressing Body Image Issues While Teaching Academic Course: The Group- Theory and Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Hai College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Tel Hai Academic College
Record Dates: First submitted 2017-08-27; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Self Esteem; Body Image
Keywords: Self Esteem; Body Image; Eating disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active participants (Experimental): The first 20 students who signed up for the course: "The group- theory and practice" were included. No exclusion criteria were used. Full attendance in the course which includes 13 sessions was mandatory. In each session, students were assigned to different body image tasks that were discussed in the coming session. All students completed a self-report questionnaire at baseline and conclusion of the course.
  Interventions: Behavioral: Academic course "The group- theory and practice"
- Controls (No Intervention): All the other students, that requested to sign up for the course but did not have a place, served as control group. All students completed a self-report questionnaire at baseline and conclusion of the course.

INTERVENTIONS:
Behavioral: Academic course "The group- theory and practice" — Active participation in the course "The group- theory and practice".
  Arms: Active participants

SUMMARY:
MSc. course addressing the issue of body image among nutrition students while delivering the course "The group- theory and practice". A non-randomized controlled trial was conducted between 2014 and 2016 with 135 dietetics' students in Tel Hai Academic College, Israel. Changes in body image and eating disorders features were assessed between course conclusion and baseline among participants within controlled efficacy study.

DETAILED DESCRIPTION:
An innovative MSc. course addressing the issue of body image among nutrition students while delivering the course "The group- theory and practice". A non-randomized controlled trial was conducted between 2014 and 2016 with 135 dietetics' students in Tel Hai Academic College, Israel. All stages of the project were compliant with the Declaration of Helsinki. Informed written consent was obtained from all participants in the study. Changes in body image and eating disorders features were assessed between course conclusion and baseline among participants within controlled efficacy study.

The primary task of the described course is four folded:

1. Explore the theory and practice of key dimensions of groups and group facilitation.
2. Active participation in body image group
3. Develop deep understanding of the dynamics and processes through participants' own experience and behavior as it occurs in real time.
4. Develop ideas about how and what have been learned, that can be applied to their role as nutritionists and group facilitators.

The described course provides an alternative to the traditional psycho-education approach using an experiential and analogize approach during the course sessions. The three parts session starts with 45 minutes of frontal lecture focused on group theories. In the next 45 minutes, half of the students participate in a body image group while the other half serve as outside observers using structured forms. All participants filled the day before structured exercise, which expose them to the main issues that will be discussed and practiced in the group session. In the last 45 minutes, the observers report about their observation and the whole class discuss the group dynamics observed. The course includes 42 hours, 3 hours in each of the 14 sessions.

This model of learning emphasize deep learning of the "participant role" as well as the "facilitator role".

ELIGIBILITY:
Inclusion Criteria:

* Must be student enrolled at Tel-Hai Academic College.
* Must be among first 20 students to sign up for the course.

Exclusion Criteria:

* Non-students.
* Not among first 20 students to sign up for the course.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
The Rosenberg self-esteem questionnaire | Each participant was be assessed for a total duration of 4 months, measuring a change in rosenberg self esteem scale
  The Rosenberg self-esteem questionnaire in (Rosenberg, 1965). It contains 10 items rated on a scale ranging from 1 (strongly disagree) to 4 (strongly agree). The total score is obtained via summation with items 2,5,6,8,9 being scored oppositely. Scores on the RSE have been shown to demonstrate acceptable internal consistency, test-retest reliability over a 2-week period, and convergent validity (Robinson & Shaver, 1973)
The Body Image States Scale (BISS) | Each participant was be assessed for a total duration of 4 months, measuring a change in The Body Image States Scale
  The Body Image States Scale (BISS) (Cash, 2002). Measures persons' evaluative/affective body-image states. It is a six-item scale with acceptably internally consistent. Scoring of the BISS: The measure is the composite mean of the six 9-point items. The measure should be scored so that low scores reflect more negative body image states and high scores reflect more positive states. Prior to taking the mean of the six items, reverse score items 2, 4, and 6.
The Body Shape Questionnaire BSQ-34 | Each participant was assessed for a total duration of 4 months, measuring a change in The Body Shape Questionnaire BSQ-34
  The Body Shape Questionnaire BSQ-34 (BSQ; Cooper et al.,1986), a 34-item self-report measure of body dissatisfaction cognitions and preoccupation, consists of items rated on a frequency scale of one ("never") to six ("always") and yields a range of total scores from 34 to 204.
The Eating Disorder Inventory-2 | Each participant was assessed for a total duration of 4 months, measuring a change in The Eating Disorder Inventory-2
  The Eating Disorder Inventory-2 (EDI-2) (Garner, 1991). This self-report inventory contains 91 items divided into eleven subscales rated on a 0-4 point scoring system. 3 items are specific to eating disorders and 8 are general psychological scales that while not specific are relevant to eating disorders.
The Body Esteem Scale for Adolescents and Adults | Each participant was assessed for a total duration of 4 months, measuring a change in The Body Esteem Scale
  The Body Esteem Scale for Adolescents and Adults (BES) (Mendelson, Mendelson, & White, 2001) was used to measure self-evaluation of body appearance. A total score was computed, with higher values indicating more positive body-esteem.
The Body Appreciation Scale | Each participant was assessed for a total duration of 4 months, measuring a change in The Body Appreciation Scale
  The Body Appreciation Scale (BAS) (Avalos et al, 2005). A 13 items self-report questionnaire reflecting aspects of positive body image. Items were designed to assess the extent to which women: (a) hold favorable opinions of their bodies, (b) accept their bodies in spite of their weight, body shape, and imperfections, (c) respect their bodies by attending to their body's needs and engaging in healthy behaviors, and (d) protect their body image by rejecting unrealistic images of the thin-ideal prototype portrayed in the media. BAS items are rated along a 5-point scale (i.e., 1 = never, 2 = seldom, 3 = sometimes, 4 = often, 5 = always) and are averaged to obtain an overall body appreciation score. Higher scores reflect greater body appreciation.
Satisfaction | Each participant was assessed at the end of the intervention, for 1 day (while completing questionnaire).
  Overall satisfaction from course was rated on a scale of 1 to 5

SECONDARY OUTCOMES:
Demographic information | Each participant was assessed at baseline, for 1 day (while completing questionnaire).
  Demographic information was obtained from each participant at baseline.
Personal details: social security number, age, email address | Each participant was assessed at baseline, for 1 day (while completing questionnaire).
  Personal details were obtained from each participant at baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Hai Academic College, Kiryat Shmona, Israel

IPD SHARING:
Plan to Share IPD: No